CLINICAL TRIAL: NCT00002768
Title: AUTOLOGOUS STEM CELL TRANSPLANTATION FOR ACUTE MYELOID LEUKEMIA IN SECOND REMISSION: A PHASE II STUDY
Brief Title: Chemotherapy Plus Peripheral Stem Cell Transplantation in Treating Patients With Acute Myeloid Leukemia in Second Remission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-9620; U10CA031946 (NIH); CLB-9620; CDR0000064734 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2004-04-22 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia in remission; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute promyelocytic leukemia (M3); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute megakaryoblastic leukemia (M7); adult acute monocytic leukemia (M5b); adult acute minimally differentiated myeloid leukemia (M0)
MeSH Terms: conditions — Leukemia; Leukemia, Erythroblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Busulfan; Cytarabine; Etoposide; Methotrexate; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous stem cell transplantation (Experimental): Patients receive consolidation chemotherapy followed by autologous stem cell transplantation
  Interventions: Biological: filgrastim; Drug: busulfan; Drug: cytarabine; Drug: etoposide; Drug: methotrexate; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim — 10 microgram/kg body wt subcutaneously daily beginning on d 14 and con't until peripheral blood collection is completed
  Other Names: G-CSF
Drug: busulfan — 1 mg/kg PO q 6 hrs for 16 doses on days -7 thru -4.
Drug: cytarabine — 2000 mg/ sq meter IV over 2 hours q 12 hrs x 8 doses on days 1-4
  Other Names: Ara-C
Drug: etoposide — 40 mg/kg (total dose) IV cont infusion over 96 hrs on days 1-4 of consolidation therapy and 60 mg/kg IV over 4 hrs on day -3 of transplant
Drug: methotrexate — For patients with documented CNS disease at first relapse, 12 mg intrathecal for a total of 6 doses given before and/or after transplantation
Procedure: peripheral blood stem cell transplantation — Infusion on Day 0

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of peripheral stem cell transplantation following chemotherapy in treating patients with acute myeloid leukemia in second remission.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the ability of mobilization using cytarabine, etoposide, and filgrastim (G-CSF), conditioning using busulfan and etoposide, and autologous peripheral blood stem cell transplantation to generate a 2-year disease-free survival rate in at least 30% of patients with acute myeloid leukemia (AML) in second complete remission. II. Determine whether the treatment-related mortality can be limited to less than 20% in patients treated with this regimen. III. Determine whether adequate numbers of PBSC can be collected in these patients. IV. Determine the engraftment kinetics of primed PBSC obtained from these patients.

OUTLINE: Mobilization/harvest: Patients receive cytarabine IV over 2 hours every 12 hours and etoposide IV continuously on days 1-4. Filgrastim (G-CSF) is administered subcutaneously (SC) beginning on day 14 and continuing until peripheral blood stem cells (PBSC) are harvested. When blood counts recover, PBSC are harvested and selected for CD34+ cells. Conditioning: Beginning at least 4 weeks after hospital discharge for mobilization and harvest and when blood counts recover, patients receive oral busulfan every 6 hours on days -7 to -4 and etoposide IV over 4 hours on day -3. PBSC are reinfused on day 0. G-CSF is administered SC beginning on day 0 and continuing until blood counts recover. Patients with documented CNS disease at first relapse receive methotrexate intrathecally at intervals of 1 week or greater before and/or after PBSC transplantation for a total of 6 doses. Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 26-48 patients will be accrued within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of acute myeloid leukemia (AML) in second complete remission (CR) for 30 days to less than 1 year before study entry Second CR defined by the following: Neutrophil count at least 1,000/mm3 Platelet count at least 100,000/mm3 Normal bone marrow morphology with no excess blasts (greater than 5%) No myelodysplasia No extramedullary or CNS leukemia Initial diagnosis of de novo AML (M0-M7) No prior myelodysplasia No myeloproliferative disease No secondary AML Cytogenetics not required No cytogenetic evidence of persistent leukemia if cytogenetics performed

PATIENT CHARACTERISTICS: Age: 15 to 69 Hematopoietic: See Disease Characteristics Granulocyte count at least 1,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL AST less than 3 times normal Alkaline phosphatase less than 3 times normal No cirrhosis or chronic hepatitis Biopsy required if chronic liver disease suspected (history of alcohol abuse or possible hepatitis) Renal: Creatinine less than 2.0 mg/dL Other: Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior bone marrow/stem cell transplantation Chemotherapy: Prior non-ablative chemotherapy at initial diagnosis, during initial remission, or as reinduction therapy (to produce current second remission) allowed At least 4 weeks since hospital discharge after reinduction therapy Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: No prior post-remission therapy for second remission

Ages: 15 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 1996-06; Primary Completion 2003-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles Linker, MD, Study Chair — University of California, San Francisco
Locations (3):
- United States (3):
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey

REFERENCES:
- [Result] Linker CA, Owzar K, Powell B, Hurd D, Damon LE, Archer LE, Larson RA; Cancer and Leukemia Group B. Auto-SCT for AML in second remission: CALGB study 9620. Bone Marrow Transplant. 2009 Sep;44(6):353-9. doi: 10.1038/bmt.2009.36. Epub 2009 Mar 16. PMID 19289999